CLINICAL TRIAL: NCT02129075
Title: A Phase II, Open-Label, Multicenter, Randomized Study of CDX-1401, a Dendritic Cell Targeting NY-ESO-1 Vaccine, in Patients With Malignant Melanoma Pre-Treated With Recombinant CDX-301, a Recombinant Human Flt3 Ligand
Brief Title: A Vaccine (CDX-1401) With or Without a Biologic Drug (CDX-301) for the Treatment of Patients With Stage IIB-IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00898; NCI-2014-00898 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CITN-07-FLT3L; CITN-07-FLT3L (Other: Cancer Immunotherapy Trials Network); CITN-07-FLT3L (Other: CTEP); P30CA015704 (NIH); U01CA154967 (NIH)
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Cutaneous Melanoma; Melanoma; Melanoma of Unknown Primary; Mucosal Melanoma; Ocular Melanoma; Stage IIB Cutaneous Melanoma AJCC v6 and v7; Stage IIC Cutaneous Melanoma AJCC v6 and v7; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — poly ICLC; flt3 ligand protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (CDX-301, CDX-1401, poly-ICLC) (Experimental): Patients receive recombinant Flt3 ligand (CDX-301) SC on days -7 to -1, 1-3, and 22-28 of cycle 1 and only on days 1-3 of cycle 2. Patients also receive CDX-1401 SC or ID on day 1 of each cycle and poly-ICLC SC on days 1-2 of each cycle. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Drug: Poly ICLC; Biological: Recombinant Flt3 Ligand
- Arm II (CDX-1401, poly-ICLC) (Active Comparator): Patients receive CDX-1401 and poly-ICLC as in Arm I. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Drug: Poly ICLC

INTERVENTIONS:
Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401 — Given SC or ID
  Other Names: CDX-1401
Drug: Poly ICLC — Given SC
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid
Biological: Recombinant Flt3 Ligand — Given SC
  Other Names: CDX-301; FLT 3 Ligand; FLT3 Ligand; Flt3-Ligand; Flt3L; Mobist; Mobista; rhuFlt3L
  Arms: Arm I (CDX-301, CDX-1401, poly-ICLC)

SUMMARY:
This phase II trial studies the effect of a vaccine called CDX-1401 given with or without a biologic drug called CDX-301 in treating patients with stage IIB-IV melanoma. The cancer vaccine CDX-1401 attaches to a protein that is made in tumor cells. The vaccine helps the body recognize the tumor to fight the cancer. The biologic drug CDX-301 may help the body make more of the tumor fighting cells, known as dendritic cells. Another biologic drug, poly-ICLC, may stimulate the immune system and help these dendritic cells mature so that they can recognize the tumor. Giving CDX-301 may make the immune response to a combination of CDX-1401 and poly-ICLC better.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether the immune response to NY-ESO-1 elicited by vaccination with DEC-205/NY-ESO-1 fusion protein CDX-1401 (CDX-1401) plus polyinosinic-polycytidylic acid stabilized with poly-L-lysine and carboxymethylcellulose (poly-ICLC) is substantially increased by prior expansion in the number of circulating dendritic cells (DC) by therapy with recombinant Flt3 ligand (CDX-301) (fms-related tyrosine kinase 3 ligand [Flt3L]).

SECONDARY OBJECTIVES:

I. To assess the effect of the vaccine regimen on immune responses to other ongoing and nascent antitumor response antigens associated with melanoma (e.g., PRAME, MAGE-A3, p53, and gp100) as well as memory viral responses (influenza A) and chronic viral responses (cytomegalovirus [CMV], Epstein-Barr virus [EBV]).

II. To assess the effect of the vaccine regimen on the frequency and phenotypic character of peripheral blood mononuclear cell (PBMC) subsets including DCs, monocyte populations, T cells, and natural killer (NK) cells.

III. To assess the safety, tolerability, and clinical efficacy of the vaccine regimens.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive recombinant Flt3 ligand (CDX-301) subcutaneously (SC) on days -7 to -1, 1-3, and 22-28 of cycle 1 and only on days 1-3 of cycle 2. Patients also receive CDX-1401 SC or intradermally (ID) on day 1 of each cycle and poly-ICLC SC on days 1-2 of each cycle. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive CDX-1401 and poly-ICLC as in Arm I. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 and 12 weeks and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fully resected stage IIb through IV melanoma, with melanoma validated by histology or cytology, who have NOT received prior therapy.

  * Patients may have had primary cutaneous, mucosal, or ocular melanoma or metastasis from an unknown primary site.
  * Tissue should be submitted for evaluation of NY-ESO-1 expression and T-cell infiltrates. However, availability of tissue and/or positivity for NY-ESO-1 is not mandatory.
* Prior radiation, chemotherapy or biologics NOT allowed
* Not currently receiving any anticancer therapy
* Age >= 18 years

  * Because no dosing or adverse event (AE) data are currently available on the use of CDX-1401 or CDX-301 in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-1
* Life expectancy of at least 6 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Hemoglobin > 9 g/dL
* Total bilirubin < 1.5 x institutional upper limit of normal (bilirubin < 3 x institutional upper limit of normal for Gilbert's syndrome)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine < 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The first six patients enrolled in the Flt3L arm of the study cannot be human immunodeficiency virus (HIV)-positive. After the evaluation of safety in the first 6 patients, HIV-positive patients with adequate immune function as evidenced by stable CD4 counts >= 350/mm^3 are allowed to participate if the following criteria are met:

  * maintained on stable antiretroviral therapy with no significant drug interactions, and
  * no recent history of acquired immunodeficiency syndrome (AIDS) indicator conditions (> 2 years from enrolling in trial), and
  * physician providing patient's care for HIV must also approve of patient entering the study
* Females of childbearing potential must have a negative pregnancy test within 7 days before the initiation of protocol therapy.

  * The effects of CDX-1401 or CDX-301 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) before study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception before the study, for the duration of study participation, and 4 months after completion of CDX-1401 or CDX-301 administration.
  * NOTE: Subjects are considered not of child-bearing potential if they are surgically sterile, they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy, or they are postmenopausal. Menopause is the age associated with complete cessation of menstrual cycles, menses, and implies the loss of reproductive potential. By a practical definition, it assumes menopause after 1 year without menses with an appropriate clinical profile at the appropriate age.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had cytotoxic chemotherapy, radiotherapy, interferon (IFN), or ipilimumab before entering the study
* Immunosuppressive therapy within 30 days prior to initiation of protocol therapy
* Steroid therapy, or steroid therapy with more than 7 consecutive days of steroids within the prior 4 weeks

  * The use of prednisone or equivalent < 0.125 mg/kg/day (absolute maximum of 10 mg/day) as replacement therapy is permitted
  * Inhaled or topical corticosteroids are permitted
* Patients who are receiving any other investigational agents
* Current or history of systemic autoimmune disease requiring systemic therapy.

  * NOTE: The following will not be exclusionary:

    * The presence of laboratory evidence of autoimmune disease (e.g., positive antinuclear antibody [ANA] titer) without associated symptoms
    * Clinical evidence of vitiligo
    * Other forms of depigmenting illness
* Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association Class III or IV), active angina pectoris, or recent myocardial infarction (within the last 6 months)
* Cirrhosis or chronic hepatitis C virus positivity or chronic hepatitis B infection

  * NOTE: A positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B virus surface antibody [HBsAb]-positive and hepatitis B virus core antibody [HBcAb]-negative), or a fully resolved acute hepatitis B virus infection is not an exclusion criterion
* Known history of immunodeficiency disorder other than HIV-positive status
* Extensive active brain disease including symptomatic brain metastases or presence of leptomeningeal disease

  * NOTE: Patients with brain metastasis, after definitive therapy with surgery or stereotactic radiation and stable off steroids for >= 4 weeks, are eligible
* Other invasive cancers that are clinically active
* Pregnancy or nursing or unwilling to take adequate birth control during therapy

  * NOTE: Pregnant women are excluded from this study because CDX-1401 or CDX-301 and poly-ICLC have an unknown potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CDX-1401 or CDX-301, breastfeeding should be discontinued if the mother is treated with CDX-1401 or CDX-301 and poly-ICLC
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CDX-1401 or CDX-301 or poly-ICLC
* Prior organ allograft or allogeneic transplantation, if the transplanted tissue is still in place
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Medical or psychiatric illness that would, in the opinion of the investigator, preclude participation in the study or the ability of patients to provide informed consent for themselves
* History of pulmonary disease such as emphysema or chronic obstructive pulmonary disease (COPD) (forced expiratory volume in 1 second [FEV1] < 60% of predicted for height and age). Pulmonary function tests (PFTs) are required in patients with prolonged smoking history or symptoms of respiratory dysfunction
* Vaccinations other than those given as part of this research study (with the exception of influenza vaccine) are prohibited throughout the duration of study participation.

  * NOTE: Influenza vaccination (inactivated) is permitted during the flu season. The preferred time is 7 to 14 days after CDX-1401 administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2016-03-28 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (7):
- United States (7):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Bhardwaj N, Friedlander PA, Pavlick AC, Ernstoff MS, Gastman BR, Hanks BA, Curti BD, Albertini MR, Luke JJ, Blazquez AB, Balan S, Bedognetti D, Beechem JM, Crocker AS, D'Amico L, Danaher P, Davis TA, Hawthorne T, Hess BW, Keler T, Lundgren L, Morishima C, Ramchurren N, Rinchai D, Salazar AM, Salim BA, Sharon E, Vitale LA, Wang E, Warren S, Yellin MJ, Disis ML, Cheever MA, Fling SP. Flt3 ligand augments immune responses to anti-DEC-205-NY-ESO-1 vaccine through expansion of dendritic cell subsets. Nat Cancer. 2020 Dec;1(12):1204-1217. doi: 10.1038/s43018-020-00143-y. Epub 2020 Nov 16. PMID 35121932

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No enrolled participants were excluded from the study before assignment to groups.
Groups:
- Arm I (CDX-301, CDX-1401, and Poly-ICLC): Patients receive recombinant flt3 ligand (CDX-301) SC on days -7 to -1, 1-3, and 22-28 of course 1 and on days 1-3 of course 2 only; DEC-205/NY-ESO-1 fusion protein CDX-1401 SC or ID on days 1 and 2; and poly-ICLC SC on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  DEC-205/NY-ESO-1 Fusion Protein CDX-1401: Given SC or ID
  Laboratory Biomarker Analysis: Correlative studies
  Neoantigen-based Melanoma-Poly-ICLC Vaccine: Given SC
  Pharmacological Study: Correlative studies
  Recombinant Flt3 Ligand: Given SC
- Arm II (CDX-1401 and Poly-ICLC): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401and poly-ICLC as in Arm I. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  DEC-205/NY-ESO-1 Fusion Protein CDX-1401: Given SC or ID
  Laboratory Biomarker Analysis: Correlative studies
  Neoantigen-based Melanoma-Poly-ICLC Vaccine: Given SC
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Arm I (CDX-301, CDX-1401, and Poly-ICLC) | Arm II (CDX-1401 and Poly-ICLC)
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (CDX-301, CDX-1401, and Poly-ICLC) | Arm II (CDX-1401 and Poly-ICLC) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 25 | 47
  >=65 years | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (13.4) | 51.6 (14.5) | 53.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 28 | 58
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 30 | 28 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Immune T-cell Response to NY-ESO-1
Description: Response rates will be analyzed by tabulating the frequency of positive response for each assay by antigen and treatment arm at each time point for which an assessment is performed. Response rates will be presented with their corresponding 95% confidence interval estimates calculated using the score test method. Fisher's exact tests will be used to compare cohort 1 and cohort 2 at the peak time point, with a significant difference declared if the 1-sided P value is =< 0.10.
Time Frame: At 12 weeks after final vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (CDX-301, CDX-1401, and Poly-ICLC) | Arm II (CDX-1401 and Poly-ICLC)
Number analyzed (Participants) | 28 | 26
Participants | 15 | 10

2. Secondary Outcome: T Cell Responses to Other Ongoing and Nascent Antitumor Response Antigens Associated With Melanoma (e.g. PRAME, MAGE-A3, p53, and gp1000) as Well as Memory and Chronic Viral Responses (CMV, EBV)
Description: as for outcome 1
Time Frame: Up to 12 weeks after final vaccination
Population: T cell responses to MAGE-A3 and PRAME; positive at any timepoint
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (CDX-301, CDX-1401, and Poly-ICLC): Patients receive recombinant flt3 ligand SC on days -7 to -1, 1-3, and 22-28 of course 1 and on days 1-3 of course 2 only; DEC-205/NY-ESO-1 fusion protein CDX-1401 SC or ID on days 1 and 2; and poly-ICLC SC on day 1. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  DEC-205/NY-ESO-1 Fusion Protein CDX-1401: Given SC or ID
  Laboratory Biomarker Analysis: Correlative studies
  Neoantigen-based Melanoma-Poly-ICLC Vaccine: Given SC
  Pharmacological Study: Correlative studies
  Recombinant Flt3 Ligand: Given SC
Arm/Group | Arm I (CDX-301, CDX-1401, and Poly-ICLC) | Arm II (CDX-1401 and Poly-ICLC)
Number analyzed (Participants) | 30 | 28
Participants | 7 | 7

3. Secondary Outcome: Frequency and Phenotypic Character of PBMC Subsets Including DCs, Monocyte Populations, T Cells, and NK Cells - Highest Peak Fold Change Over Baseline (Log 2 Fold)
Description: Graphical and tabular summaries of the assay data will be made. Linear mixed effects model and possibly weighted generalized estimating equation methods will be considered for a supportive analysis of the longitudinal data over time.
Time Frame: Up to 12 weeks after final vaccination
Population: Only a subset of patient specimens were needed to meet statistical power. 15 participants were analyzed in Arm I (CDX-301, CDX-1401, and poly-ICLC and 16 participants were analyzed in Arm II (CDX-1401 and poly-ICLC). One less patient in Arm 1 was analyzed due to sample quality.
Measure: Mean (Standard Deviation); unit: log 2 fold change
Arm/Group | Arm I (CDX-301, CDX-1401, and Poly-ICLC) | Arm II (CDX-1401 and Poly-ICLC)
Number analyzed (Participants) | 15 | 16
log 2 fold change
  cDCs | 30.4 (16.98) | 0.9 (0.26)
  Monocytes | 6.1 (2.11) | 1.0 (0.18)
  CD4 T cells | 1.2 (0.28) | 1.1 (0.27)
  NK CD56br cells | 5.8 (2.84) | 1.26 (0.32)
  CD8 T cells | 1.3 (0.36) | 1.0 (.26)
  pDC | 16.5 (7.27) | 0.8 (0.24)

4. Secondary Outcome: Tumor Recurrence
Description: Time to first recurrence from first vaccine among subjects who have experienced recurrence. (days)
Time Frame: Up to 600 days from first vaccine
Population: Analysis is reported for the number of subjects with recurrence (N=12 Arm I) (N=9 Arm II)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I (CDX-301, CDX-1401, and Poly-ICLC) | Arm II (CDX-1401 and Poly-ICLC)
Number analyzed (Participants) | 12 | 9
days | 360.3 (191.1) | 389.2 (223.2)

5. Secondary Outcome: Overall Survival
Description: Overall survival not assessed
Time Frame: Up to 1 year after patient's 12 week visit
Population: Data not collected
Arm/Group | Arm I (CDX-301, CDX-1401, and Poly-ICLC) | Arm II (CDX-1401 and Poly-ICLC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Systematic evaluation by clinicaltrials.gov definition
Arm/Group | Arm I (CDX-301, CDX-1401, and Poly-ICLC) | Arm II (CDX-1401 and Poly-ICLC)
Serious Adverse Events (participants affected / at risk) | 0/30 | 4/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (CDX-301, CDX-1401, and Poly-ICLC) (N=30) | Arm II (CDX-1401 and Poly-ICLC) (N=30)
General disorders and administration site conditions (General disorders) | 0 (0) | 1 (1)
Infections and infestations (Infections and infestations) | NA | 1 (1)
Nervous system disorders (Nervous system disorders) | NA | 1 (1)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | NA | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (CDX-301, CDX-1401, and Poly-ICLC) (N=30) | Arm II (CDX-1401 and Poly-ICLC) (N=30)
General disorders and administration site conditions (General disorders) | 30 (509) | 30 (322) — Injection site reactions
Nervous system disorders (Nervous system disorders) | 17 (35) | 19 (49)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 20 (56) | 18 (33)
Gastrointestinal disorders (Gastrointestinal disorders) | 15 (37) | 17 (44)
Investigations (Investigations) | 14 (43) | 14 (49)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 15 (21) | 14 (24)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 15 (51) | 12 (28)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 13 (27) | 13 (24)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 13 (30) | 10 (17)
Infections and infestations (Infections and infestations) | 7 (10) | 9 (12)
Vascular disorders (Vascular disorders) | 8 (20) | 6 (26)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 10 (10) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 6 (8) | 4 (4)
Eye disorders (Eye disorders) | 4 (6) | 3 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Renal and urinary disorders (Renal and urinary disorders) | 2 (2) | 3 (4)
Cardiac disorders (Cardiac disorders) | 1 (2) | 2 (2)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 2 (2)
Immune system disorders (Immune system disorders) | 0 (0) | 1 (1)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less